CLINICAL TRIAL: NCT00259181
Title: Examination of the Immersion of Provisional Crown Material in Chlorhexidine Gluconate on Dental Plaque Formation in Vivo
Brief Title: A Protocol for the Use of Chlorhexidine Gluconate Saturation for the Reduction of Dental Biofilm Formation on Polymethylmethacrylate Restoration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 191058HMO-CTIL
Record Dates: First submitted 2005-11-24; First posted 2005-11-29 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2007-12

CONDITIONS: Dental Plaque
Keywords: chlorhexidine gluconate; polymethylmethacrylate; Anti-Bacterial Agents
MeSH Terms: conditions — Dental Plaque

INTERVENTIONS:
Procedure: saturation of polymethylmethacrylate with chlorhexidine gluconate to reduce in vivo plaque formation

SUMMARY:
Chlorhexidine gluconate (CHX), as an anti plaque agent, is commonly used with a variety of products. In this study we, the investigators at Hadassah Medical Organization, intend to examine the efficacy of a single dip in CHX of provisional restoration prior to oral cementation. If the protocol is effective, we intend to calibrate it and recommend clinical use of the protocol. The examination of biofilm formation will be both with electron microscope and confocal scanning laser microscope.

ELIGIBILITY:
Inclusion Criteria:

* Any volunteer without systemic condition

Exclusion Criteria:

* Intake of antibiotic drug three months prior to experiment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Start 2005-01

PRIMARY OUTCOMES:
calibration of a preventative protocol for biofilm formation measured by confocal scanning laser microscope and scanning electron microscope

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Perez Davidi, DMD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- See also: Michael Perez Davidi — http://www.mypd.co.il